CLINICAL TRIAL: NCT07296887
Title: Implement and Evaluate the CARE Tool in a Randomized Trial
Brief Title: CARE Tool Study Aim 3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-x479; U19CA291430 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Cancer; Prostate Cancer; Lung Cancer; Colorectal Cancer
Keywords: Insurance; Insurance coverage; Cancer; Cost of medical care; Financial toxicity
MeSH Terms: conditions — Prostatic Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Neoplasms; Financial Stress | interventions — Quality Indicators, Health Care

STUDY DESIGN:
Intervention Model Description: Patient participants will be randomized to one of two arms, the CARE Tool or standard financial education information, and participate in surveys. Participants enrolled as site staff and members of the care team will complete a training on the CARE Tool and participate in surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Patients - Care Tool (Intervention) (Experimental): Patients will review the web-based CARE Tool after enrollment. Patients will complete a survey immediately after reviewing the website and a 3 month follow-up survey.
  Interventions: Other: CARE Tool
- Arm 2: Patients - Standard of care financial education information (Control) (Active Comparator): Patients will review standard web-based financial education information after enrollment. Patients will complete a survey immediately after reviewing the website and a 3 month follow up survey.
  Interventions: Other: Financial education information
- Arm 3: Implementation champions - CARE training (Experimental): Participants who are members of the care team and have been identified as implementation champions will complete training on the CARE Tool and cost conversations. Participants will complete a survey after the training and a post-recruitment survey at the end of the trial.
  Interventions: Other: CARE Tool Training

INTERVENTIONS:
Other: Financial education information — Standard financial education resources will be provided to patients enrolled in the control arm. Financial education will be accessible via website and provided by the participating site.
  Arms: Arm 2: Patients - Standard of care financial education information (Control)
Other: CARE Tool — The CARE Tool is a web-based tool provided to patients after enrollment. The CARE Tool provides patients with individualized information about cancer care costs, health insurance, and resources to assist with costs.
  Arms: Arm 1: Patients - Care Tool (Intervention)
Other: CARE Tool Training — Members of the care team who have been identified as implementation champions will undergo training on cost conversations, how to use the CARE Tool, and how to implement the CARE Tool in their clinical workflow.
  Arms: Arm 3: Implementation champions - CARE training

SUMMARY:
This study is a multi-site randomized trial to study the implementation of the CARE Tool and evaluate the CARE Tool. The CARE Tool is a web-based tool that gives people information about cancer care costs, health insurance, and resources to help with costs. Overall, the study aims to help patients with cancer overcome barriers they face navigating insurance and accessing financial resources.

ELIGIBILITY:
Inclusion Criteria for Implementation champions:

- Members of the cancer care team (e.g., physicians, nurses, research coordinators, financial navigators, social workers) that work with patients receiving treatment for gynecologic, lung, prostate, or colorectal cancer; or members of the billing team and employee of Siteman Cancer Center, Barnes Jewish Hospital, Washington University, Delbert Day Cancer Institute at Phelps Health, or Alton Memorial Hospital

Exclusion Criteria for Implementation champions:

* Implementation champions are ineligible if they are non-employees of Siteman Cancer Center, Barnes Jewish Hospital, Washington University, Delbert Day Cancer Institute at Phelps Health, or Alton Memorial Hospital
* Do not treat patients for gynecologic, prostate, lung, or colorectal cancer

Inclusion Criteria for Patients:

* Age 18 and over
* Primary or recurrent diagnosis of gynecologic, prostate, lung, or colorectal cancer in the last 12 months
* Receiving cancer treatment from Siteman Cancer Center, Delbert Day Cancer Institute at Phelps Health, or Alton Memorial Hospital
* Self-reported ability to read and speak English

Exclusion Criteria for Patients:

* Under the age of 18
* Not diagnosed with gynecologic, prostate, lung, or colorectal cancer within the previous 12 months from recruitment
* Not receiving care at Siteman Cancer Center, Delbert Day Cancer Institute at Phelps Health, or Alton Memorial Hospital
* Cannot give consent due to cognitive or emotional barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient's comprehensive score for financial toxicity (COST) | Completion of initial survey to completion of follow up survey (total estimated time is 3 months)
  COST will be calculated by the sum of 11-items according to the validated measure. The items are scored on a 5-point Likert scale as follows: 0-Not at all, 1-A little bit, 2-Somewhat, 3-Quite a bit, and 4-Very much. Total possible range is 0-44 and the lower the score indicates greater financial toxicity. Scores will be summarized using means and 95% confidence intervals. Changes between timepoints will be analyzed by a two-sample t-test.
Patient's score of self-efficacy for communicating about care costs measured with the Decision Self-Efficacy Scale | Completion of initial survey to completion of follow up survey (total estimated time is 3 months)
  The measure of self-efficacy for communicating about care costs is adapted from the validated tool Decision Self-Efficacy Scale. The Decision Self-Efficacy Scale measures self-confidence or belief in one's abilities in decision making, including shared decision making. Three-items from the Decision Self-Efficacy Scale will be used to measure self-efficacy for communicating about care costs. The three items will be measured by a 3-point Likert scale as follows: 0-Not Confident, 2-A Little Confident, and 4-A lot confident. A higher score indicates greater self-efficacy in decision making. The total score will be calculated according to the validated measure. Scores will be summarized using means and 95% confidence intervals. Changes between timepoints will be analyzed by a two-sample t-test.
Patient's health insurance literacy measure (HILM) score | Completion of initial survey to completion of follow up survey (total estimated time is 3 months)
  HILM score is calculated from a 6-item questionnaire according to the validated measure. Each item is measured by a 4-point Likert scale as follows: 1-Not at all confident, 2-Slightly confident, 3-Moderately confident, and 4-Very confident. Total possible range is 0-100 where 0 represents the lowest possible health insurance literacy level (more difficulty navigating insurance) and 100 represents the highest (more confidence in choosing/using insurance). Scores will be summarized using means and 95% confidence intervals. Changes between timepoints will be analyzed by a two-sample t-test.

SECONDARY OUTCOMES:
Patient's reported adherence to therapy & delayed care | Completion of initial survey to completion of follow up survey (total estimated time is 3 months)
  Patient reported delayed care will be calculated from responses to three-items adapted from the National Health Interview Survey (NHIS). The three items have four categorical answers: Yes, No, I don't know, and Prefer not to answer. Scores will be summarized using frequencies. Changes between timepoints will be analyzed using sample proportions and 95% Clopper-Pearson Confidence Intervals. Changes between timepoints will be analyzed by a Pearson Chi-square test. .
Feasibility of Intervention Measure (FIM) - Adapted | At start of recruitment and at completion recruitment (total estimated time is 2 years)
  FIM will be assessed by implementation champions' response to a single item from the FIM measure on the initial and follow up survey. FIM is measured by a 5-point Likert scale: 1-Completely disagree, 2-Disagree, 3-Neither agree nor Disagree, 4-Agree, or 5-Completely agree. A higher score indicates greater feasibility of the intervention in practice. Outcome will be summarized using means and 95% confidence intervals. Changes between surveys will be analyzed by a two-sample t-test.
Acceptability of Intervention Measure (AIM) - Adapted | At start of recruitment and at completion recruitment (total estimated time is 2 years)
  AIM will be assessed by implementation champions' response to a single item from the AIM measure on the initial and follow up survey. AIM is measured by a 5-point Likert scale: 1-Completely disagree, 2-Disagree, 3-Neither agree nor Disagree, 4-Agree, or 5-Completely agree. A higher score indicates greater acceptability by subjects of the intervention. Outcome will be summarized using means and 95% confidence intervals. Changes between surveys will be analyzed by a two-sample t-test.
Intervention Appropriateness Measure (IAM) - Adapted | At start of recruitment and at completion recruitment (total estimated time is 2 years)
  IAM will be assessed by implementation champions' response to a single item from the IAM measure on the initial and follow up survey. IAM is measured by a 5-point Likert scale: 1-Completely disagree, 2-Disagree, 3-Neither agree nor Disagree, 4-Agree, or 5-Completely agree. A higher score indicates greater appropriateness of the intervention. Outcome will be summarized using means and 95% confidence intervals. Changes between surveys will be analyzed by a two-sample t-test.

OTHER OUTCOMES:
Organizational Readiness-Adapted | At start of recruitment and at completion recruitment (total estimated time is 2 years)
  Organizational readiness will be assessed by implementation champions' response to 6 items adapted from the MORE measure for organizational readiness and 3 items adapted from the organizational readiness for implementing change (ORIC) measure. MORE items are measured on a 4-point Likert scale: 1-Not willing, 2-Somewhat willing, 3-Willing, and 4-Very willing. A higher score indicates greater organizational readiness. ORIC items are measured on a 5-point Likert scale: 1-Disagree, 2-Somewhat Disagree, 3-Neither agree nor Disagree, 4-Somewhat Agree, or 5-Agree. A higher score indicates greater organizational readiness to implement change. Changes between surveys will be analyzed by a two-sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Housten, OTD, MSCI, OTR/L, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Alton Memorial Hospital, Alton, Illinois
  - Delbert Day Cancer Institute at Phelps Health, Rolla, Missouri
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Participants can share their data for future research. Data such as age, sex, gender identity, race, and ethnicity, will be redacted to strip identifiers and minimize risks of unauthorized disclosure of personal identifiers.
  Common data elements (CDEs), identified by NCI and the ACCERT sites, will include identifiable information like zip code and county. Data from this optional survey could identify participants and may be shared with the NCI and ACCERT study teams .
  Publicly available documentation will include the study protocol, survey questions, codebook, univariate statistics, and study-level metadata. The codebook will include a description of each variable with the question number and text, variable name, variable label, value labels, and standard codes for missing values-including codes for non-applicable, "don't know," or prefer not to answer. We may share algorithms produced for analysis of CDEs.
  Users must agree to the conditions of use governing access to the data.
Supporting Information: Study Protocol
Time Frame: Final submission and deposit of the study data will occur at the end of data collection. Study data deposited will be available to the research community in perpetuity. Datasets underlying methodological publications will be shared at or prior to initial publication date.
Access Criteria: Researchers within the ACCERT consortium and those who provide a methodologically sound plan.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu